CLINICAL TRIAL: NCT03538223
Title: Music Listening to Reduce Anxiety and Stress in Patients Undergoing Radiotherapy
Brief Title: Music Listening in Radiotherapy Treatment
Acronym: MuLi_RT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Collaborators: University of Pavia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2179 CE
Record Dates: First submitted 2018-04-26; First posted 2018-05-29 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Breast Cancer
Keywords: Music listening; Radiotherapy; Breast cancer; Psychological rehabilitation
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Radioterapy+"Melomics-Health" Listening (Experimental): The musical content is composed by an algorithm (named "Melomics-Health") with the purpose of acting psychologically and physiologically on the person: the music follows a constant, melodic trend with a reduced musical density; time is unchanged and there are no significant dynamic and tonal variations. Patients will undergo to music listening for 15 minutes (5 tracks lasting 3 minutes each) before radiotherapy session. Appropriate earphones will be used in order to focus their attention on the musical-sound component and to isolate themselves from the external context.
  Interventions: Other: Music Listening; Radiation: Radiotherapy
- Radiotherapy+Individualized Listening (Experimental): The musical content is based on the patient's preferred music (chosen by patients with the support of the music therapist) with the purpose of acting psychologically and physiologically on the person. Patients will undergo to music listening for 15 minutes before radiotherapy session. Appropriate earphones will be used in order to focus their attention on the musical-sound component and to isolate themselves from the external context.
  Interventions: Other: Music Listening; Radiation: Radiotherapy
- Radiotherapy+No Music Listening (Other): Patients will undergo the standard treatment (radiotherapy) without music support.
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Other: Music Listening — Participants will undergo two different types of music before radiotherapy sessions
  Arms: Radioterapy+"Melomics-Health" Listening; Radiotherapy+Individualized Listening
Radiation: Radiotherapy — All participants will undergo radiotherapy according to breast cancer post surgery protocol

SUMMARY:
Music and music therapy are now widely used as non-pharmacological intervention techniques in different clinical and therapeutic settings.

The present study includes the use of musical listening related to the concept of "Music Medicine", a possibility of modifying the psycho-physiological state of the patient through the targeted use of musical pieces respondent to specific parameters and musical structures able to interact in particular conditions with the psycho-somatic imbalances to which the person is subjected.

In particular, in this study, in addition to proposing a traditional listening method, the music used in one of the research arms will be composed of an artificial intelligence called "Melomics-Health".

The objective of the study is to verify whether the perception of anxiety and stress in cancer patients undergoing Radiotherapy is influenced by music listening ("Melomics-Health" music vs listening to favorite music). Sixty breast cancer surgical patients, candidates for post-operative radiotherapy with a healing purpose. Patients who will undergo Radiation therapy for the first time in their lives will be included.

Patients will be recruited in this randomized controlled study with a sequential enrollment and, in the case of inclusion, will be assigned to one of the following 3 groups: a) "Melomics-Health" music listening group (n = 20); b) favorite music listening group (n = 20); c) no-music control group (n = 20). Music groups will undergo 15 minutes music listening immediately before the simulation and the first 5 sessions of radiotherapy.

Patients will be subjected to a psychological assessment focused on anxiety (State-Trait Anxiety Inventory) and distress (Psychological Distress Inventory) dimensions at the baseline (T0), at the end of the treatments (T1) and at the Follow-up (T2, 2 weeks after the fifth session of Radiotherapy). A specific questionnaire will also be submitted to the patients included in music groups. This questionnaire will allow the music therapist to acquire specific qualitative information regarding the different types of music listening and the responses of the subjects to them.

Descriptive statistics will be produced for all the variables detected.The effectiveness of musical listening in relation to the psychological aspects considered will be evaluated by applying analysis of variance models.

DETAILED DESCRIPTION:
Introduction: Music and music therapy are now widely used as non-pharmacological intervention techniques in different clinical and therapeutic settings.

Scientific literature includes a large number of studies structured according to scientific criteria and its presence is documented by the existence of numerous systematic reviews about this topic (including Cochrane Reviews). Some of these reviews, together with single studies, concern to the use of music in the hospital setting in different areas as: the pre-surgical and surgical phases, specific oncology interventions and also radiotherapy / chemiotherapy treatments. In these contexts the applicative experiences are generally characterized by two factors: the music therapy technique used that is the use of musical listening rather than active music therapy interventions (interaction between patient and therapist through musical instruments) and the possible effectiveness of music on momentary symptoms as anxiety, stress and pain deriving from illness conditions and / or from particularly invasive medical procedures.

The present study includes the use of musical listening related to the concept of "Music Medicine", a possibility of modifying the psycho-physiological state of the patient through the targeted use of musical pieces respondent to specific parameters and musical structures able to interact in particular conditions (such as illness, surgery, etc) with the psycho-somatic imbalances to which the person is subjected. On the other hand, it has been demonstrated that music can also significantly affect vital parameters and neurochemical processes leading to significant modifications of these aspects.

In particular, in this study, in addition to proposing a traditional listening method, the music used in one of the research arms will be composed of an artificial intelligence called "Melomics-Health" and created in collaboration with the Research Group in Biomimetics of the University of Malaga. This way of composing music gives the possibility to intervene on the design of the music itself, creating the necessary conditions for its use in the therapeutic field. Music can be composed on the basis of specific sound parameters and appropriate musical structures with the aim of achieving the intended therapeutic objective. In this direction, numerous studies have been undertaken whose initial results are really encouraging. One of the advantages of this technology is given by the possibility of forging and shaping the music according to the therapeutic objective, leaving to the artificial intelligence the task to produce it. This perspective represents an absolute innovation and creates considerable potentialities in the use of music listening aimed at the care and health of the individual. The concept above exposed concerning the action of sound and music on the individual together with the use of "Melomics-Health" technology, create the necessary conditions for the fulfillment of the proposed study.

Material and Methods: Sixty breast cancer surgical patients, candidates for post-operative radiotherapy with a healing purpose.

Study design: patients will be recruited in this randomized controlled study with a sequential enrollment and, in the case of inclusion, will be assigned to one of the following 3 groups: a) music listening group (n = 20) (with "Melomics-Health" music) created in relation to the objective of the study; b) favorite music listening group (n = 20) (who will listen to a play-list created with the collaboration of a music therapist; c) a control group (n = 20) to which no musical listening will be proposed. A randomization list, in accordance with a completely randomized parallel group study design, will be generated at the beginning of the study. Within the randomization list, each subject will be uniquely identified by a numerical code that will allow its identification during the entire duration of the study if necessary. Patient identification data will be kept in a separate and properly protected database. The type of intervention expected for this study does not allow its blind conducting for the investigator and for the participant. However, the blindness of psychological and statistical evaluations will be guaranteed in order to reduce the possibility of distortions due to observer or statistical biases.

Assessment: patients will be subjected to a psychological assessment focused on anxiety and distress dimensions correlated to the planned medical procedure and more generally to the clinical condition. At the time of patients enrollment (screening) a clinical / anamnestic assessment will be performed, the inclusion criteria will be verified and appropriate patients will be asked to sign the informed consent. At the baseline (T0), at the end of the treatments (T1) and at the Follow-up (T2, 2 weeks after the fifth session of Radiotherapy) the State-Trait Anxiety Inventory form Y (STAI) and the Psychological Distress Inventory (PDI) will be administered. At T1 phase (conclusion of the treatments) a specific questionnaire will also be submitted to the patients of groups A and B. This questionnaire will allow the music therapist to acquire specific qualitative information regarding the different types of music listening and the responses of the subjects to them.

Procedures: Phase 1. The staff identified by the research team, having verified the presence of inclusion criteria, will consider the patient enrollment and will assign it to one of the treatment arms ("Melomics-Health" listening, individualized listening and absence of music) on the basis of the Principal Investigator indications who manages the randomization list. The patient will be initially explained the motivations and general contents of the study. Only after the patient's effective adherence to the treatment and after the signing of the informed consent, the procedure of the study will be shown the patient according to the assignment group. Patients who adhere to the proposal will be asked to provide some personal information and will subsequently be subjected to the assessments expected by the study. Any failure in obtaining the informed consent or any case of refusal to the request to participate in the study by the enrolled patient, will make it consider as a drop-out patient.

Phase 2. Before the simulation session the psychological scales expected at T0 will be submitted to the patients (STAI of state and of trait and Psychological Distress Inventory - PDI). The treatments will be repeated during the simulation session and for the first five sessions of Radiotherapy. During the last day of treatment (T1, 5th session) and 2 weeks after the conclusion of the treatments (T2) all patients will be evaluated again through the administration of STAI of state and of trait and Psychological Distress Inventory - PDI. During the last day of treatment, a specific musical questionnaire will also be submitted to patients in groups A and B.

Statistics: A statistical analysis plan will be defined in detail before the start of the data analysis phase, taking into account the exploratory nature of the study. In general, descriptive statistics will be produced for all the variables detected. The effectiveness of musical listening in relation to the psychological aspects considered will be evaluated by applying the appropriate models of analysis of variance. All randomized patients for whom at least one available follow-up will be included in the main statistical analyzes (Intention-To-Treat population, with Last Observation Carried Forward); secondary analyzes will be carried out on the subgroup consisting only of patients who have completed the entire follow-up (Per-Protocol population).

ELIGIBILITY:
Inclusion Criteria:

* patients who will undergo Radiation therapy for the first time in their lives
* patients who are candidates for hypofractionated partial breast irradiation with a duration of at least 10 sessions
* patients who signed the informed consent

Exclusion Criteria:

* patients with associated diseases that preclude the understanding of the study contents (eg patients with established psychiatric disorders and / or with significant cognitive deficits)
* patients with significant hearing loss
* patients already previously subjected to music therapy or therapy based on music listening
* patients with musical skills (musical training or musical practice> 3 years).
* patients who are candidates for hypofractionated partial breast irradiation with a duration equal to or less than 10 sessions

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Women with breast cancer
Enrollment: 60 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Anxiety reduction | Baseline (T0) vs 2 weeks (T1, i.e. end of radiotherapy treatment)
  Difference in State-Trait Anxiety Inventory (STAI) score. There are 2 subscales within this measure: 1) the State Anxiety Scale (S-Anxiety) evaluating the current state of anxiety; 2) the Trait Anxiety Scale (T-Anxiety) evaluating relatively stable aspects of "anxiety proneness". Range of scores for each subtest is 20-80, the higher score indicating greater anxiety.

SECONDARY OUTCOMES:
Anxiety reduction | Baseline (T0) vs 4 weeks (T2, two weeks after the end of radiotherapy treatment)
  Difference in State-Trait Anxiety Inventory (STAI) score. There are 2 subscales within this measure: 1) the State Anxiety Scale (S-Anxiety) evaluating the current state of anxiety; 2) the Trait Anxiety Scale (T-Anxiety) evaluating relatively stable aspects of "anxiety proneness". Range of scores for each subtest is 20-80, the higher score indicating greater anxiety.
Stress reduction | Baseline (T0) vs 2 weeks (T1, i.e. end of radiotherapy treatment)
  Difference in Psychological Distress Inventory (PDI) score. Score range is from 13 (low distress level) to 65 (high distress level).
Stress reduction | Baseline (T0) vs 4 weeks (T2, two weeks after the end of radiotherapy treatment)
  Difference in Psychological Distress Inventory (PDI) score. Score range is from 13 (low distress level) to 65 (high distress level).

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Raglio, PhD, Principal Investigator — Istituti Clinici Scientifici Maugeri SpA
Locations (1):
- Istituti Clinici Scientifici Maugeri SpA, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bradt J, Dileo C, Magill L, Teague A. Music interventions for improving psychological and physical outcomes in cancer patients. Cochrane Database Syst Rev. 2016 Aug 15;(8):CD006911. doi: 10.1002/14651858.CD006911.pub3. PMID 27524661
- [Background] Bradt J, Dileo C, Shim M. Music interventions for preoperative anxiety. Cochrane Database Syst Rev. 2013 Jun 6;2013(6):CD006908. doi: 10.1002/14651858.CD006908.pub2. PMID 23740695
- [Background] Chen LC, Wang TF, Shih YN, Wu LJ. Fifteen-minute music intervention reduces pre-radiotherapy anxiety in oncology patients. Eur J Oncol Nurs. 2013 Aug;17(4):436-41. doi: 10.1016/j.ejon.2012.11.002. Epub 2012 Dec 4. PMID 23218591
- [Background] Clark M, Isaacks-Downton G, Wells N, Redlin-Frazier S, Eck C, Hepworth JT, Chakravarthy B. Use of preferred music to reduce emotional distress and symptom activity during radiation therapy. J Music Ther. 2006 Fall;43(3):247-65. doi: 10.1093/jmt/43.3.247. PMID 17037953
- [Background] Morasso G, Costantini M, Baracco G, Borreani C, Capelli M. Assessing psychological distress in cancer patients: validation of a self-administered questionnaire. Oncology. 1996 Jul-Aug;53(4):295-302. doi: 10.1159/000227576. PMID 8692533
- [Background] O'Callaghan C, Sproston M, Wilkinson K, Willis D, Milner A, Grocke D, Wheeler G. Effect of self-selected music on adults' anxiety and subjective experiences during initial radiotherapy treatment: a randomised controlled trial and qualitative research. J Med Imaging Radiat Oncol. 2012 Aug;56(4):473-7. doi: 10.1111/j.1754-9485.2012.02395.x. Epub 2012 May 28. PMID 22883658
- [Background] Raglio A, Vico F. Music and Technology: The Curative Algorithm. Front Psychol. 2017 Nov 24;8:2055. doi: 10.3389/fpsyg.2017.02055. eCollection 2017. No abstract available. PMID 29250008
- [Background] Rossetti A, Chadha M, Torres BN, Lee JK, Hylton D, Loewy JV, Harrison LB. The Impact of Music Therapy on Anxiety in Cancer Patients Undergoing Simulation for Radiation Therapy. Int J Radiat Oncol Biol Phys. 2017 Sep 1;99(1):103-110. doi: 10.1016/j.ijrobp.2017.05.003. Epub 2017 May 8. PMID 28816136
- [Result] Raglio A, Oddone E, Meaglia I, Monti MC, Gnesi M, Gontero G, Imbriani C, Ivaldi GB. Conventional and Algorithmic Music Listening before Radiotherapy Treatment: A Randomized Controlled Pilot Study. Brain Sci. 2021 Dec 8;11(12):1618. doi: 10.3390/brainsci11121618. PMID 34942921